CLINICAL TRIAL: NCT01066494
Title: A Phase IIa Pharmacokinetic and Efficacy Study of Amonafide L-malate (AS1413) in Combination With Cytarabine in Adult Patients With Acute Myeloid Leukemia (AML)
Brief Title: A Pharmacokinetic and Efficacy Study of Amonafide L-malate (AS1413) in Combination With Cytarabine in Patients With Acute Myeloid Leukemia (AML)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Antisoma Research (Industry)
Responsible Party: Fredrik Erlandsson, Antisoma
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AS1413-C-101
Record Dates: First submitted 2010-02-09; First posted 2010-02-10 (Estimated); Last update posted 2011-01-17 (Estimated); Status verified 2011-01

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML; Pgp; MDR; sAML; AS1413; Amonafide
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — amonafide; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single-arm (Experimental): Amonafide 600 mg/m2 IV over 4 hours daily on days 1-5 in combination with cytarabine 200 mg/m2 IV continuous infusion (CI) daily on days 1-7
  Interventions: Drug: Amonafide + cytarabine

INTERVENTIONS:
Drug: Amonafide + cytarabine — Amonafide 600 mg/m2 IV over 4 hours daily on days 1-5 in combination with cytarabine 200 mg/m2 IV continuous infusion (CI) daily on days 1-7

SUMMARY:
A phase IIa study to evaluate the pharmacokinetic and efficacy of amonafide L-malate (AS1413) in combination with cytarabine in treating patients with acute myeloid leukemia (AML)

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent
2. In the opinion of the Investigator able to comply with the study assessments and follow-up
3. New diagnosis of AML (i.e. >20 % blasts) as defined by the World Health Organization (WHO) classification (Vardiman 2009) or relapsed or refractory AML as defined by the persistence or recurrence of >5% blasts in bone marrow or peripheral blood following treatment.
4. ECOG Performance status ≤ 2
5. Age > 18 years and ≤ 70 years
6. Adequate hepatic function as evidenced by the following laboratory tests:

   1. Total serum bilirubin ≤ 1.5 x ULN or direct (conjugated) bilirubin ≤ 1.5 ULN unless attributable to suspected hepatic involvement with AML
   2. Serum AST and ALT ≤ 1.5 x ULN unless attributable to suspected hepatic involvement with AML
7. Adequate renal function as evidenced by serum creatinine ≤ 1.5 x ULN
8. Women of childbearing potential must have a negative serum pregnancy test. A woman of childbearing potential is defined as one who is biologically capable of becoming pregnant. This includes women who are using contraceptives or whose sexual partners are either sterile or using contraceptives
9. Left Ventricular Ejection Fraction (LVEF) > 50%, as determined by multiplegated acquisition scan (MUGA) or echocardiogram (ECHO) within 28 days prior to administration of 1st dose of remission induction chemotherapy

Exclusion Criteria:

1. Unwilling to accept the required per protocol blood and urine sample collection
2. An initial diagnosis of acute promyelocytic leukemia as defined by French- American-British criteria (Bennett 1976) (otherwise known as FAB M3)
3. Clinically active CNS leukemia
4. History of clinically significant allergic reactions attributed to compounds of similar chemical or biological composition to amonafide or cytarabine
5. Pregnant or breast feeding
6. Known HIV positive
7. Known active hepatitis B or C, or any other active liver disease
8. Evidence of pulmonary infection. Patients with evidence of pulmonary infection on screening chest x-ray should have chest computed tomography (CT) prior to starting remission induction therapy to confirm absence or presence of pulmonary infection.
9. Any major surgery or radiation therapy within 30 days prior to study entry
10. Previously received treatment with amonafide
11. Treatment with other investigational agents for any reason within 30 days prior to study entry
12. Prior remission induction therapy for AML within 30 days of starting amonafide therapy
13. Persistent non-hematologic toxicity (other than alopecia) greater than Grade 2 from prior therapy for MDS or AML
14. Serious concomitant illnesses (for example, unstable angina or myocardial infarction or stroke within 3 months prior to study entry, congestive heart

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-09 (Estimated); Study Completion 2011-01 (Estimated)

PRIMARY OUTCOMES:
To define the plasma PK Profile of amonafide and metabolite(s) | 1 year
To deine the urniary excretion of amonafide and metabolite(s) | 1 year
To investigate the fecal excretion of amonafide and metabolite(s) in selected patients | 1 year
To evaluate the safety and tolerability of amonafide in combination with cytarabine | 1 year
To evaluate the remission rate | 1 year

SECONDARY OUTCOMES:
All outcomes are of equal weighting | 1 year

CONTACTS AND LOCATIONS:
Locations (6):
- Georgia (3):
  - Institute of Haematology and Transfusiology, Tbilisi
  - Medulla - Chemotherapy and Immunotherapy Clinic, Tbilisi
  - Hema - Haematology and Chemotherapy Clinic, Tbilisi
- Ukraine (3):
  - Institure of URgent adn Recovery Surgery n.a. V.K. gusaka of Academy Medical Science of Ukraine, Donetsk
  - Kyiv bone Marrow Transplantation Centre, Kiev
  - Vinnytsya Regional clinical Hospital, Vinnytsia